CLINICAL TRIAL: NCT04436289
Title: Home Link: Post Hospital Care to Reduce HIV Mortality in South Africa
Acronym: HomeLink
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Witwatersrand, South Africa (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00214009; 5R34MH118998 (NIH)
Record Dates: First submitted 2020-06-15; First posted 2020-06-18 (Actual); Results first posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: HIV/AIDS
Keywords: home-based; post-hospital care
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to care as usual or Home Link arm. We will perform individual randomization blocked by HIV-status to enroll 30 HIV-uninfected per arm and 90 PWH per arm.
Who Masked: Investigator
Masking Description: Participants and members of the research team recruiting and implementing the strategy will be unmasked to randomization assignment due to the behavioral nature of the strategy and need for team members to explain the study arm procedures to participants. Study assignments will be masked to the investigators until all outcome data have been collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PLWH care-as-usual (CAU) study arm (No Intervention): Participants living with HIV will receive standard discharge care as provided at Tshepong Hospital during the study. This currently includes discharge counseling from a trained discharge counselor and will be provided with a follow-up return date (usually two weeks post-hospital). Discharge counseling will include a review of discharge medications and instructions regarding follow-up care visits.
- PLWH Home Link study arm (Experimental): The Home Link intervention will be delivered by a home visit team including a primary care nurse and counselor trained in patient-centered counseling. A rotating hospital-based doctor will be available for pre-home visit clinical file review and post-visit discussion, via cell phone, for decision making and input on patient care during a household visit. We have termed this individual a "discharge officer". The discharge officer will be a Tshepong clinician who is working in the hospital. Supporting Home Link is expected to take <30 minutes of the physician's time during the day. For study-specific concerns, the team will consult with a GCP-trained, PHRU research doctor based at Tshepong Hospital.
  Interventions: Behavioral: Home Link
- PLWOH care-as-usual (CAU) study arm (No Intervention): Participants living without HIV will receive standard discharge care as provided at Tshepong Hospital during the study. This currently includes discharge counseling from a trained discharge counselor and will be provided with a follow-up return date (usually two weeks post-hospital). Discharge counseling will include a review of discharge medications and instructions regarding follow-up care visits.
- PLWOH Home Link study arm (Experimental): The Home Link intervention will be delivered by a home visit team including a primary care nurse and counselor trained in patient-centered counseling. A rotating hospital-based doctor will be available for pre-home visit clinical file review and post-visit discussion, via cell phone, for decision making and input on patient care during a household visit. We have termed this individual a "discharge officer". The discharge officer will be a Tshepong clinician who is working in the hospital. Supporting Home Link is expected to take <30 minutes of the physician's time during the day. For study-specific concerns, the team will consult with a GCP-trained, PHRU research doctor based at Tshepong Hospital.
  Interventions: Behavioral: Home Link

INTERVENTIONS:
Behavioral: Home Link — In the Home Link intervention, a team will conduct home visits to (1) provide a structured clinical assessment; (2) reconcile medications, (3) provide psychosocial support through patient-centered counseling, and (4) assess home needs (food security). These visits will start one week after discharge and be repeated every two weeks until the participant is stabilized and ready to initiate lower intensity clinic-based services or three months have elapsed.
  Arms: PLWH Home Link study arm; PLWOH Home Link study arm

SUMMARY:
Background: This is a pilot randomized clinical trial (RCT) to demonstrate the feasibility and acceptability of a structural and behavioral intervention to reduce mortality following hospital discharge for people with HIV (PWH) in South Africa. Investigators' prior study showed that among 121 PWH discharged, 54% were readmitted and 26% had died by six months following discharge. In the prior study, investigators identified that missing clinic visits after discharge was associated with death. Here investigators are seeking to overcome key barriers in piloting a home-based post-hospital care intervention. Investigators' approach is informed by a conceptual model of key barriers to the care transition along with a behavioral explanatory model, the Behavioral Model for Vulnerable Populations.

The overarching goal of this study is to tailor and pilot the intervention that shifts initial post-discharge care from the out-patient clinic to the home and provides patient-centered counseling (Home Link intervention). For the intervention to prove effective it will need to substantially reduce post-discharge mortality. Specifically, in the Home Link intervention, a team will conduct home visits to (1) provide a structured clinical assessment; (2) reconcile medications, (3) provide psychosocial support through patient-centered counseling, and (4) assess home needs (food security). These visits will start one week after discharge and be repeated every two weeks until the participant is stabilized and ready to initiate lower intensity clinic-based services or three months have elapsed.

Aims: The aims of the study are to pilot a randomized clinical trial of home delivery of health services during the post-hospital period for PWH.

Methods: This project is a pilot randomized clinical trial (RCT) to refine and test the feasibility, acceptability, and preliminary effectiveness of the HomeLink intervention. At the conclusion of the R34 grant period investigators will have a protocol and procedural manual ready for a full RCT powered for effectiveness.

Significance: The proposed study is consistent with NIH HIV/AIDS highest priority research and the South African National Strategic Plan on HIV, tuberculosis (TB), and sexually transmitted infections (STIs) 2017-2022. The research addresses the HIV/AIDS Research Priority of "retention and engagement in these services, and achievement and maintenance of optimal prevention and treatment responses."

DETAILED DESCRIPTION:
BACKGROUND

Sub-Saharan Africa HIV mortality:

In 2016 in South Africa approximately 154,000 PWH died. Of these deaths, 110,000 have been characterized as excess mortality due to HIV (HIV associated deaths). Overall, HIV-associated deaths are associated advanced disease defined by a low cluster of differentiation 4 (CD4) count.

In-Hospital and Post-Hospital Mortality in Africa:

Inpatient mortality among people with HIV (PWH) in Africa is uniformly high ranging from 17.2 to 29.6% across the continent, including in South Africa. Following discharge from an index hospitalization the mortality is also high. In investigators' preliminary work investigators have observed a 26% mortality in the 6 months after hospital discharge. This observation is consistent with mortality from other reports: 50% mortality at twelve months and 30% and 31% at six months reported from Tanzania, Kenya, and South Africa, respectively.

Contribution of Post-Hospital Mortality to Overall Death among People with HIV:

In South Africa there are approximately 84,633 public sector acute care hospital beds of which approximately 25% are adult medicine beds. By extrapolating the post-discharge mortality investigators observed to all discharges among PWH in South Africa investigators can estimate the annual mortality among PWH with a hospital discharge in the past six months. Considering the national proportion of all admissions that are for PWH, the average length of stay, and the annual readmission rate an estimated 240,000 PWH are admitted to medicine wards in South Africa annually. A six-month post-hospital mortality of 26% suggests a total of 62,374 post-hospital deaths among PWH. This number of deaths represents 40% of the approximately 154,000 total annual deaths among PWH in South Africa. A modest reduction in post-hospital deaths could substantially reduce overall HIV mortality in South Africa.

Causes of Post-Hospital Death:

Some post-hospital deaths may be unavoidable due to advanced or incurable disease. Other post-hospital deaths may be avoidable with improved retention in care. A study from Johannesburg, South Africa assessed loss from care for HIV-TB co-infected patients; only 42% of patients discharged were known to have been to an HIV clinic within 30 days of hospital discharge [the time needed to obtain or refill antiretroviral therapy (ART) prescriptions at the time of the study]. Similarly in Investigators' preliminary study, only 19% of participants attended a scheduled follow-up visit. Failure to attend a scheduled visit was associated with subsequent mortality in Investigators' preliminary study and in a report from Tanzania. At present, there is limited research regarding approaches to retaining PWH in care during the post-hospital transition.

STUDY OBJECTIVES

The overarching goal of this proposal is to demonstrate clinical trial feasibility, acceptability, and preliminary efficacy of structured post-discharge medical home visits to reduce mortality following the transition from the hospital to home. Investigators are proposing a pilot randomized clinical trial (RCT) to determine preliminary efficacy, feasibility of trial implementation and intervention delivery, acceptability of the intervention, the effect of the intervention on barriers to care, and to obtain detailed baseline psychosocial and medical needs to inform intervention refinement and explain outcomes.

The primary objectives of this study are:

1. To estimate 6 month mortality rates and assess for evidence of efficacy of the Home Link intervention compared to care as usual.
2. To determine the feasibility, acceptability, and effect of the Home Link intervention on identified barriers to care.
3. To characterize medical and behavioral needs among participants in the study.

The secondary objectives of this study are:

1. Determine post-hospital health care out-of-pocket costs for participants
2. Assess re-admission
3. Estimate 12 month mortality by study arm

SIGNIFICANCE

This study fits with the South African National Strategic Plan to increase effective HIV treatment. The study is also consistent with NIH HIV/AIDS highest priority research and the South African National Strategic Plan on HIV, TB, and STIs 2017-2022. Given the high post-discharge mortality findings from this study could contribute to approaches to reduce mortality for PWH.

METHODS

Study design:

This is a pilot randomized clinical trial (RCT) to refine and test the feasibility, acceptability, and preliminary effectiveness of Home Link.

Study setting:

This pilot operational research study will be conducted in Matlosana. All participants will be recruited from Tshepong Hospital. Eligibility will include residing within Matlosana sub-district.

Tshepong Hospital: Tshepong Hospital is a tertiary care hospital in Matlosana. An average of 30 patients are admitted to medicine wards daily. Nearly 50% are PWH.

Description of the geographical areas of study implementation:

The proposed study will be conducted at the 500 bed Tshepong Hospital in the Northwest Province. Tshepong Hospital is one of 5 hospitals in Kenneth Kaunda District and the single tertiary care public hospital serving the population of 400,000 in Matlosana. This hospital was selected due to its size, heterogeneous catchment area (rural to urban), and long-standing working relationships with the research team. Tshepong Hospital currently provides discharge services that include (1) discharge counseling and education provided by counselors and (2) a medical record notebook with a discharge summary for the patient to take to his or her clinic visits.

Rationale for selecting geographical areas of study implementation:

Investigators selected Tshepong Hospital based on a long-standing working relationship between the PI, the Perinatal HIV Research Unit (PHRU), and the Tshepong Hospital. This has included a prior study of post-hospital outcomes.

Study Population:

The study population is comprised of adults (≥18 years old), either male or female, spending at least two nights in a medical ward of Tshepong Hospital. Investigators will only include individuals with known HIV status, either HIV-positive or HIV-negative. Investigators propose to recruit up to 180 HIV-positive and 60 HIV-uninfected participants. Randomization to the intervention vs control arms will be stratified by HIV status.

Pre-discharge study procedures:

All participants will have a baseline demographic health and psychosocial questionnaire (E001, E002).

Care-as-usual (CAU) study arm:

Participants will receive standard discharge care as provided at Tshepong Hospital during the study. This currently includes discharge counseling from a trained discharge counselor and will be provided with a follow-up return date (usually two weeks post-hospital). Discharge counseling will include a review of discharge medications and instructions regarding follow-up care visits.

Home Link study arm:

The Home Link intervention will be delivered by a home visit team including a primary care nurse and counselor trained in patient-centered. A rotating hospital-based doctor will be available for pre-home visit clinical file review and post-visit discussion, via cell phone, for decision making and input on patient care during a household visit. Investigators have termed this individual a "discharge officer". The discharge officer will be a Tshepong clinician who is working in the hospital. Supporting Home Link is expected to take <30 minutes of the physician's time during the day. For study-specific concerns, the team will consult with a Good Clinical Practice (GCP)-trained, PHRU research doctor based at the Tshepong Hospital.

Post-discharge follow-up:

The primary outcome is mortality six months after hospital discharge. Secondary outcomes include mortality 12 months after hospital discharge, number of nights spent in a hospital, number of ambulatory clinical encounters after the index hospitalization, and patient out-of-pocket costs for medical care. Outcomes will be assessed through scheduled contact and completion of a structured questionnaire with the participant or designated next of kin (either telephonic or in person if telephonic fails) at 8, 12, 26, and 52 weeks. Mortality will be further ascertained through a 26 and 52 week review of the Tshepong Hospital file (including the affiliated Klerksdorp hospital files) and matching of participant national identification numbers to the vital statistics register through consultation with the Department of Home Affairs. Repeat hospitalization will be ascertained using self-report / next of kin report and hospital records. Most subsequent hospitalizations can be expected to be at Tshepong Hospital due to the substantial distance to reach the next nearest hospital (>50 km to a lower level facility). In Investigators' prior experience investigators have observed rare use of alternative hospitals. Clinic visit data will be ascertained by self-report followed by verification through review of clinic paper or electronic (tier.net) records and National Health Laboratory Service electronic records (TrackCare).

ELIGIBILITY:
Inclusion Criteria:

* Tested for HIV (can be living with HIV or HIV-uninfected)
* Residing within Matlosana sub-district
* Agree to post-discharge follow-up including home visit
* Able to provide informed consent or, if lacking capacity at the time of recruitment (if unable to answer basic orientation questions including name, month/year, and residence location), as determined by the study team, having a next of kin able to provide informed consent

Exclusion Criteria:

* <18 years of age
* Length of stay <2 nights
* Unknown HIV status at the point of study screening and enrollment
* Failure by the patient or next of kin to provide informed consent to be followed up by study staff after discharge
* Residing outside of Matlosana sub-district
* Not speaking any of the languages spoken by the study team

Late exclusions occurring after enrollment:

* Death prior to hospital discharge
* Discharged too late for the study team to deliver the intervention
* Transfer to another hospital
* Relocation outside of Matlosana sub-district at the point of discharge or within 7 days of discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hoffmann, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Tshepong Hospital, Klerksdorp, North West, South Africa

IPD SHARING:
Plan to Share IPD: Yes
De-identified trial data will be made available one year after completion of all study activities.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: One year after completion of study activities.
Access Criteria: Contact PI.

RESULTS

PARTICIPANT FLOW:
Groups:
- PLWH Care-as-usual (CAU) Study Arm; PLWOH Care as Usual (CAU) Study Arm: Participants will receive standard discharge care as provided at Tshepong Hospital during the study. This currently includes discharge counseling from a trained discharge counselor and will be provided with a follow-up return date (usually two weeks post-hospital). Discharge counseling will include a review of discharge medications and instructions regarding follow-up care visits.
Period: Overall Study
Arm/Group | PLWH Home Link Study Arm | PLWH Care-as-usual (CAU) Study Arm | PLWOH Home Link Study Arm | PLWOH Care as Usual (CAU) Study Arm
Started | 63 | 62 | 35 | 35
Completed | 55 | 51 | 30 | 31
Not Completed | 8 | 11 | 5 | 4
Not completed — Death prior to hospital discharge | 8 | 5 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 4 | 0
Not completed — Extended hospital stay | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 4 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Analysis population excludes those who were late exclusions from the primary trial due to death prior to discharge or an extended hospital stay
Groups:
- PLWOH Care-as-usual (CAU) Study Arm: Participants will receive standard discharge care as provided at Tshepong Hospital during the study. This currently includes discharge counseling from a trained discharge counselor and will be provided with a follow-up return date (usually two weeks post-hospital). Discharge counseling will include a review of discharge medications and instructions regarding follow-up care visits.
- Total: Total of all reporting groups
Arm/Group | PLWH Home Link Study Arm | PLWH Care-as-usual (CAU) Study Arm | PLWOH Home Link Study Arm | PLWOH Care-as-usual (CAU) Study Arm | Total
Number analyzed (Participants) | 55 | 56 | 35 | 34 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 53 | 54 | 29 | 29 | 165
  >=65 years | 2 | 2 | 6 | 5 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 37 | 19 | 20 | 116
  Male | 15 | 19 | 16 | 14 | 64
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 55 | 56 | 35 | 34 | 180
HIV status at admission [Count of Participants; unit: Participants]
  HIV-negative | 0 | 0 | 35 | 34 | 69
  HIV-positive without reported prior knowledge | 3 | 2 | 0 | 0 | 5
  Known HIV-positive on admission | 52 | 54 | 0 | 0 | 106
Advanced HIV at admission [Count of Participants; unit: Participants]
  No | 13 | 19 | 0 | 0 | 32
  Yes | 41 | 37 | 0 | 0 | 78
  N/A - HIV negative | 0 | 0 | 35 | 34 | 69
  Missing | 1 | 0 | 0 | 0 | 1
On ART at admission [Count of Participants; unit: Participants]
  No | 26 | 15 | 0 | 0 | 41
  Yes | 28 | 41 | 0 | 0 | 69
  Missing | 1 | 0 | 0 | 0 | 1
  N/A - HIV negative | 0 | 0 | 35 | 34 | 69
Most recent CD4 count (result within the last 6 months) [Count of Participants; unit: Participants]
  <50 | 14 | 13 | 0 | 0 | 27
  50-199 | 16 | 12 | 0 | 0 | 28
  200-349 | 6 | 7 | 0 | 0 | 13
  350-499 | 9 | 13 | 0 | 0 | 22
  Missing | 10 | 11 | 0 | 0 | 21
  N/A - HIV negative | 0 | 0 | 35 | 34 | 69
Viral load result [Count of Participants; unit: Participants]
  <50 | 7 | 19 | 0 | 0 | 26
  050-999 | 13 | 13 | 0 | 0 | 26
  1000+ | 35 | 23 | 0 | 0 | 58
  Missing | 0 | 1 | 0 | 0 | 1
  N/A - HIV negative | 0 | 0 | 35 | 34 | 69
Food security [Count of Participants; unit: Participants]
  Food secure | 22 | 47 | 20 | 31 | 120
  Food insecure | 33 | 9 | 15 | 3 | 60
Alcohol use [Count of Participants; unit: Participants]
  Never | 30 | 42 | 24 | 22 | 118
  Monthly or less | 12 | 9 | 9 | 9 | 39
  2-4 per month | 4 | 1 | 1 | 3 | 9
  2-3 per week | 2 | 0 | 1 | 0 | 3
  4 or more per week | 7 | 4 | 0 | 0 | 11
HIV stigma scale [Median (Inter-Quartile Range); unit: units on a scale] — HIV stigma scale refers to the "12-item HIV stigma scale". Response options were 'strongly agree', 'agree', 'disagree', and 'strongly disagree'. Strongly agree was coded as 4 points, agree was 3 points, disagree was 2 points, and strongly disagree was coded as 1 point. The total score was calculated by summing the responses to all 12 questions for each participant. The minimum possible score is 12 and the maximum possible score is 48. A higher total score indicates greater stigma. Population: HIV stigma scale was assessed for participants living with HIV only. Data not collected from participants living without HIV
  units on a scale
    number analyzed (Participants) | 55 | 56 | 0 | 0 | 111
    (all) | 22 [17 to 27] | 21 [17.5 to 24] |  |  | 21 [17 to 26]
Modified social support (scaled score) [Median (Inter-Quartile Range); unit: scaled score] — 8-question "Modified Medical Outcomes Study (MOS) Social Support scale" - responses were 'always' (5 points), 'often' (4 points), 'sometimes' (3 points), 'rarely' (2 points), and 'never' (1 point). Total score was calculated by summing responses to all 8 questions for each participant. Min possible score is 8 (7 for 1 participant missing 1 question) and max possible score is 40 (35 for 1 participant missing 1 question). The score was then scaled using the following calculation: 100*((total score - min score)/(max score - min score)). A higher scaled score indicated greater social support.
  scaled score | 100 [87.5 to 100] | 100 [93.75 to 100] | 100 [75 to 100] | 100 [87.5 to 100] | 100 [87.5 to 100]
CES-D 10 [Median (Inter-Quartile Range); unit: units on a scale] — 10-question Centre for Epidemiologic Studies Depression Scale. Response options: rarely or none of the time, some of or a little of the time, a moderate/medium amount of time, and most of the time. Rarely coded as 0 points, some of the time as 1 point, moderate/medium as 2 points, most of the time as 3 points, except for questions 5 and 8 which are reverse coded. Total score calculated by summing responses to all 10 questions for each participant. Min possible score is 0 and the max possible score is 30 (note 2 participants missing 1 question each). Score >10 indicated evidence of depression.
  units on a scale | 5 [3 to 9] | 6 [4 to 8] | 6 [3 to 11] | 5 [4 to 8] | 6 [4 to 9]
Duration of hospitalization [Median (Inter-Quartile Range); unit: days] — Population: Two participants were missing records for the index admission. Thus duration of index hospitalization available for 178 of 180 participants.
  days
    number analyzed (Participants) | 54 | 56 | 35 | 33 | 178
    (all) | 7 [3 to 12] | 6 [3 to 12] | 4 [3 to 6] | 6 [3 to 9] | 6 [3 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Mortality at 6 Months
Description: Number of deaths from any cause.
Time Frame: 6 months after hospital discharge
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PLWH Home Link Study Arm | PLWH Care-as-usual (CAU) Study Arm | PLWOH Home Link Study Arm | PLWOH Care-as-usual (CAU) Study Arm
Number analyzed (Participants) | 55 | 56 | 35 | 34
Participants | 4 | 10 | 3 | 4

2. Secondary Outcome: Mortality at 12 Months
Description: Number of deaths from any cause.
Time Frame: 12 months after hospital discharge
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PLWH Home Link Study Arm | PLWH Care-as-usual (CAU) Study Arm | PLWOH Home Link Study Arm | PLWOH Care-as-usual (CAU) Study Arm
Number analyzed (Participants) | 55 | 56 | 35 | 34
Participants | 7 | 12 | 8 | 7

3. Secondary Outcome: Time (Days) to Any Non-acute Follow-up
Description: Time to first clinic or home visit post-hospital discharge.
Time Frame: Up to 52 weeks post-hospital discharge
Population: Among participants with at least one clinic or home visit
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | PLWH Home Link Study Arm | PLWH Care-as-usual (CAU) Study Arm | PLWOH Home Link Study Arm | PLWOH Care-as-usual (CAU) Study Arm
Number analyzed (Participants) | 53 | 45 | 32 | 25
days | 13 [11 to 19] | 28 [15 to 64] | 13 [11 to 25] | 31 [27 to 90]

4. Secondary Outcome: Number of Outpatient Follow-up Care Encounters
Description: Number of outpatient follow-up care (clinic or home visit) encounters
Time Frame: Up to 52 weeks post-hospital discharge
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: visits
Groups:
- PLWOH Home Link: The Home Link intervention will be delivered by a home visit team including a primary care nurse and counselor trained in patient-centered counseling. A rotating hospital-based doctor will be available for pre-home visit clinical file review and post-visit discussion, via cell phone, for decision making and input on patient care during a household visit. We have termed this individual a "discharge officer". The discharge officer will be a Tshepong clinician who is working in the hospital. Supporting Home Link is expected to take <30 minutes of the physician's time during the day. For study-specific concerns, the team will consult with a GCP-trained, PHRU research doctor based at Tshepong Hospital.
  Home Link: In the Home Link intervention, a team will conduct home visits to (1) provide a structured clinical assessment; (2) reconcile medications, (3) provide psychosocial support through patient-centered counseling, and (4) assess home needs (food security). These visits will start one week after discharge and be repeated every two weeks until the participant is stabilized and ready to initiate lower intensity clinic-based services or three months have elapsed.
Arm/Group | PLWH Home Link Study Arm | PLWH Care-as-usual (CAU) Study Arm | PLWOH Home Link | PLWOH Care-as-usual (CAU) Study Arm
Number analyzed (Participants) | 55 | 56 | 35 | 34
visits | 11 [7 to 14] | 3.5 [1.5 to 7] | 7 [4 to 12] | 4 [0 to 6]

5. Secondary Outcome: Number of Nights of Hospital Readmission
Description: Number of nights spent in hospital post-initial discharge (among those with at least one readmission)
Time Frame: Up to 52 weeks post-hospital discharge
Population: Among those with at least one readmission
Measure: Median (Inter-Quartile Range); unit: nights
Arm/Group | PLWH Home Link Study Arm | PLWH Care-as-usual (CAU) Study Arm | PLWOH Home Link Study Arm | PLWOH Care-as-usual (CAU) Study Arm
Number analyzed (Participants) | 21 | 24 | 17 | 12
nights | 9 [6 to 14] | 11.5 [6 to 21] | 10 [3 to 17] | 11.5 [6.5 to 20.5]

6. Secondary Outcome: Cost of Care
Description: Participant-reported out-of-pocket costs for medical care
Time Frame: Up to 52 weeks post-hospital discharge
Population: Data not collected for specific study outcome
Arm/Group | PLWH Home Link Study Arm | PLWH Care-as-usual (CAU) Study Arm | PLWOH Home Link Study Arm | PLWOH Care as Usual (CAU) Study Arm
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants Completing In-depth Interviews to Assess Acceptability of the Intervention
Description: Acceptability questionnaire and in-depth interviews with 7 acceptability domains for healthcare workers (HCWs) and participants and in-depth interviews for HCWs and participants. An a priori code book will be developed that reflects key analytic concepts of predisposing, enabling, and need characteristics from the Andersen Behavioral Model. During the process of reading and coding of transcripts using this initial coding scheme, additional codes may be added to document emerging themes of interest.
Time Frame: Up to 52 weeks post-hospital discharge
Population: Intervention arm participants who completed in-depth interviews. Care-as-usual (CAU) arm participants were not interviewed.
Measure: Number; unit: participants
Arm/Group | PLWH Home Link Study Arm | PLWH Care-as-usual (CAU) Study Arm | PLWOH Home Link Study Arm | PLWOH Care as Usual (CAU) Study Arm
Number analyzed (Participants) | 33 | 0 | 8 | 0
participants | 33 |  | 8 |

8. Secondary Outcome: Feasibility of Clinical Trial as Assessed by Enrollment Percentage
Description: Percentage of approached and eligible individuals who enroll.
Time Frame: Up to 52 weeks
Population: Among all screened participants who met eligibility criteria (pre-randomization).
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Individuals: Individuals screened for study participation who met eligibility criteria
Arm/Group | Eligible Individuals
Number analyzed (Participants) | 340
Participants | 195

9. Secondary Outcome: Feasibility of Clinical Trial as Assessed by Percentage of Participants With Complete Follow-up
Description: Feasibility of clinical trial will be determined by the percentage of participants with complete follow-up.
Time Frame: Up to 52 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PLWH Home Link Study Arm | PLWH Care-as-usual (CAU) Study Arm | PLWOH Home Link Study Arm | PLWOH Care-as-usual (CAU) Study Arm
Number analyzed (Participants) | 55 | 56 | 35 | 34
Participants | 55 | 51 | 30 | 31

10. Secondary Outcome: Feasibility of Intervention as Assessed by Participant Program Completion
Description: The number of intervention arm participants with home visit #1 completed, completion of the 12 week follow-up, and vital status ascertainment at 6 months.
Time Frame: Up to 6 months
Population: Feasibility of the intervention assessed among intervention arm participants only. This outcome not assessed among CAU participants.
Measure: Count of Participants; unit: Participants
Arm/Group | PLWH Home Link Study Arm | PLWH Care-as-usual (CAU) Study Arm | PLWOH Home Link Study Arm | PLWOH Care as Usual (CAU) Study Arm
Number analyzed (Participants) | 55 | 0 | 35 | 0
Participants | 50 |  | 27 |

ADVERSE EVENTS:
Time Frame: Up to 52 weeks post-discharge
Description: Hospital admissions were not considered an adverse event as they were a study outcome. All-cause mortality was evaluated among all randomized participants (n=195). Adverse events were evaluated among participants who were discharged from their index admission (n=180).
Arm/Group | PLWH Home Link Study Arm | PLWH Care-as-usual (CAU) Study Arm | PLWOH Home Link Study Arm | PLWOH Care-as-usual (CAU) Study Arm
All-Cause Mortality (participants affected / at risk) | 15/63 | 17/62 | 8/35 | 8/35
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/56 | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 0/55 | 0/56 | 0/35 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-03): https://cdn.clinicaltrials.gov/large-docs/89/NCT04436289/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/89/NCT04436289/ICF_001.pdf